CLINICAL TRIAL: NCT04205357
Title: Phase I Trial Combining Sulfasalazine and Gamma Knife Radiosurgery for Recurrent Glioblastoma
Brief Title: Sulfasalazine and Stereotactic Radiosurgery for Recurrent Glioblastoma
Acronym: SAS-GKRS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other); Northwell Health (Other); Weill Medical College of Cornell University (Other); University of Bergen (Other); Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2019/6834
Record Dates: First submitted 2019-11-21; First posted 2019-12-19 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Glioma; Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma | interventions — Sulfasalazine; Radiosurgery

STUDY DESIGN:
Intervention Model Description: 3 + 3 dose escalation design: Cohort 1 (3-6 patients): 1.5 gr Sulfasalazine x 1 for 3 days Cohort 2 (3-6 patients): 3.0 gr Sulfasalazine x 1 for 3 days Cohort 3 (3-6 patients): 4.5 gr SSulfasalazine x 1 for 3 days Cohort 4 (3-6 patients): 6.0 gr Sulfasalazine x 1 for 3 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sulfasalazine in addition to stereotactic radiosurgery (Other): 3 + 3 dose escalation The first cohort of 3-6 patients will receive 1.5 g Sulfasalazine daily for 3 days before single fraction stereotactic radiosurgery utilizing 12 Gy prescription dose to the tumor margin.
  The second, third and fourth cohort will receive 3 days pretreatment with 3 g, 4.5 g and 6 g Sulfasalazine, respectively, before 12 Gy single fraction stereotactic radiosurgery.
  Interventions: Drug: Sulfasalazine

INTERVENTIONS:
Drug: Sulfasalazine — Sulfasalazine combined with stereotactic radiosurgery
  Other Names: Stereotactic radiosurgery

SUMMARY:
This study evaluates the safety associated with the addition of sulfasalazine to stereotactic radiosurgery for recurrent glioblastoma. Sulfasalazine is a potential tumor selective radiosensitizer.

DETAILED DESCRIPTION:
Glioblastoma is the most aggressive and most common type of primary brain cancer. Standard treatment at diagnosis is surgery followed by high dose radiation therapy and chemotherapy. Despite initial treatment nearly all patients will experience recurrence of the tumor with a dismal prognosis. There is no consensus on standard of care at recurrence. Reoperation is associated with a high risk of complications and further conventional radiation therapy is often not possible as the maximum tolerated dose to the normal brain has already been given. In addition most tumors have developed resistance towards chemotherapy. Stereotactic radiosurgery (SRS) may be administered despite prior initial radiation treatment but in order to avoid radiation induced complications only limited doses to limited tumor volumes can be applied.

Developing new strategies to improve the effect of radiation selectively on tumor cells without simultaneously increase the radiation induced damage of normal brain would be valuable.

The investigators have shown in experimental studies that the drug sulfasalazine enhances the number of cancer cells that dies as result of radiation therapy and thereby improves survival in combination with SRS in animals with glioblastoma. Sulfasalazine inhibits the production of an antioxidant that normally protects the tumor against radiation. Hopefully the trial will result in a new and more effective treatment option for patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified glioblastoma multiforme with recurrence (first or second relapse, all subtypes) based on the Response Assessment in Neuro-Oncology criteria.
* Prior standard therapy for newly diagnosed glioblastoma consisting of surgery, standard fractionated radiotherapy to 60 Gy concomitant with Temozolomide
* Has been informed of other treatment options
* Must be eligible to gamma knife treatment
* Tumor size ≤ 3 cm in diameter (≤ 15 cm3 ) on MRI dated no more than 30 days before SRS treatment
* Must be at least 18 years of age
* Must be ambulatory with a Karnofsky performance status of ≥ 70
* Life expectancy > 12 weeks
* Laboratory parameters for vital functions should be in the normal reference range. Laboratory abnormalities that are not clinically significant are generally permitted, except for the following laboratory parameters, which must be within the ranges specified:

Hematology: White blood cell count: ≥ 3.0 x 109/l, Platelet count:: ≥ 100 x 109/l, Hemoglobin: ≥ 100 g/l, Total bilirubin level: <1.5 times the upper limit of normal (ULN) (except in patients with Gilbert's Syndrome who must have a total bilirubin less than 51,3 µmol/L), alanine aminotransferase < 3 times the ULN, Creatinine < 1.5 times the ULN, Normal prothrombin time / international normalized ratio (PT INR) < 1.4, Absolute neutrophil count: ≥ 1 x109/L without the support of filgrastim.

* More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less. Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to national/local regulations

Exclusion Criteria:

* Allergy to sulfa drugs
* Adverse reactions to salicylates
* Known hypersensitivity to sulfasalazine, its metabolites or any of the excipients (Povidone; Maize starch; magnesium stearate; colloidal silicon dioxide)
* Eligible to alternative standard treatments with temozolomide
* Treatment with sulfasalazine after glioblastoma diagnosis
* Participation in pharmacokinetic trial within 4 weeks
* Participation in immunotherapy trial within 4 weeks
* History of psychological symptoms affecting ability to consent to and/or fulfill the protocol
* Other malignant diseases and multiple sclerosis
* Pregnant or breast feeding patients.
* Porphyria
* Kidney of liver deficiencies
* Glucose-6-phosphate dehydrogenase deficiency
* Severe allergy or bronchial asthma
* History of erythema multiforme
* Significant heart failure or renal failure
* Intestinal or urinary obstruction
* Any reason why, in the opinion of the investigator, the patient should not participate (e.g. not able to comply with study procedures).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2022-10-14 (Actual)

PRIMARY OUTCOMES:
Toxicity (Common Terminology Criteria for Adverse Event v 4.0) | 1 month
  Determining the maximum tolerated and recommended dose of sulfasalazine as radiosensitizer.

SECONDARY OUTCOMES:
Intratumoral Glutathione production | 4 days
  Monitor the effect of sulfasalazine on the level of Glutathione production in glioma cells.
Presence of radiation necrosis | 1 month
  Monitor late toxicity of sulfasalazine combined with stereotactic radiosurgery on Positron Emission Tomography.
Progression free survival | 1 year
  Monitor the preliminary effect of sulfasalazine combined with stereotactic radiosurgery on local tumor control.
Overall survival | 2 years
  Assess the preliminary efficacy of sulfasalazine in combination with SRS on survival.
Quality of life (Functional Assessment of Cancer Therapy-Brain) | 1 year
  Assess the preliminary efficacy of sulfasalazine in combination with SRS on changes in quality of life utilizing the brain cancer subscale of the functional assessment of cancer therapy-Brain (FACT-Br) questionaire. The brain cancer subscale consists of twenty-three items regarding neurological concerns (range: 0-76 points). The response to the items uses a five-point scale ranging from 0 (not at all) to 4 (very much). The higher the patient score, the better the quality of life.
Karnofsky performance score (KPS) | 1 year
  Assess the preliminary efficacy of sulfasalazine in combination with stereotactic radiosurgery on changes in the Karnofsky performance score (range 0 - 100 points). The higher the score, the better is the functional performance status of the patient.
Steroid use in mg over time | 1 year
  Assess the preliminary efficacy of sulfasalazine in combination with stereotactic radiosurgery on the patients´ need for steroid medication. The change in steroid use in mg from baseline up to 1 year following radiosurgery will be evaluated using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Bente S Skeie, Principal Investigator — Haukeland University Hospial
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sleire L, Skeie BS, Netland IA, Forde HE, Dodoo E, Selheim F, Leiss L, Heggdal JI, Pedersen PH, Wang J, Enger PO. Drug repurposing: sulfasalazine sensitizes gliomas to gamma knife radiosurgery by blocking cystine uptake through system Xc-, leading to glutathione depletion. Oncogene. 2015 Dec 3;34(49):5951-9. doi: 10.1038/onc.2015.60. Epub 2015 Mar 23. PMID 25798841
- [Background] Skeie BS, Enger PO, Brogger J, Ganz JC, Thorsen F, Heggdal JI, Pedersen PH. gamma knife surgery versus reoperation for recurrent glioblastoma multiforme. World Neurosurg. 2012 Dec;78(6):658-69. doi: 10.1016/j.wneu.2012.03.024. Epub 2012 Apr 4. PMID 22484078
- [Background] Dodoo E, Huffmann B, Peredo I, Grinaker H, Sinclair G, Machinis T, Enger PO, Skeie BS, Pedersen PH, Ohlsson M, Orrego A, Kraepelien T, Barsoum P, Benmakhlouf H, Herrman L, Svensson M, Lippitz B. Increased survival using delayed gamma knife radiosurgery for recurrent high-grade glioma: a feasibility study. World Neurosurg. 2014 Nov;82(5):e623-32. doi: 10.1016/j.wneu.2014.06.011. Epub 2014 Jun 13. PMID 24930898
- [Background] Sontheimer H, Bridges RJ. Sulfasalazine for brain cancer fits. Expert Opin Investig Drugs. 2012 May;21(5):575-8. doi: 10.1517/13543784.2012.670634. Epub 2012 Mar 12. PMID 22404218
- [Background] Chung WJ, Lyons SA, Nelson GM, Hamza H, Gladson CL, Gillespie GY, Sontheimer H. Inhibition of cystine uptake disrupts the growth of primary brain tumors. J Neurosci. 2005 Aug 3;25(31):7101-10. doi: 10.1523/JNEUROSCI.5258-04.2005. PMID 16079392
- [Background] Skeie BS, Wang J, Dodoo E, Heggdal JI, Gronli J, Sleire L, Bragstad S, Ganz JC, Chekenya M, Mork S, Pedersen PH, Enger PO. Gamma knife surgery as monotherapy with clinically relevant doses prolongs survival in a human GBM xenograft model. Biomed Res Int. 2013;2013:139674. doi: 10.1155/2013/139674. Epub 2013 Nov 10. PMID 24312904
- [Background] Takeuchi S, Wada K, Nagatani K, Otani N, Osada H, Nawashiro H. Sulfasalazine and temozolomide with radiation therapy for newly diagnosed glioblastoma. Neurol India. 2014 Jan-Feb;62(1):42-7. doi: 10.4103/0028-3886.128280. PMID 24608453
- [Background] Robe PA, Martin DH, Nguyen-Khac MT, Artesi M, Deprez M, Albert A, Vanbelle S, Califice S, Bredel M, Bours V. Early termination of ISRCTN45828668, a phase 1/2 prospective, randomized study of sulfasalazine for the treatment of progressing malignant gliomas in adults. BMC Cancer. 2009 Oct 19;9:372. doi: 10.1186/1471-2407-9-372. PMID 19840379
- [Derived] Wang F, Oudaert I, Tu C, Maes A, Van der Vreken A, Vlummens P, De Bruyne E, De Veirman K, Wang Y, Fan R, Massie A, Vanderkerken K, Shang P, Menu E. System Xc- inhibition blocks bone marrow-multiple myeloma exosomal crosstalk, thereby countering bortezomib resistance. Cancer Lett. 2022 Jun 1;535:215649. doi: 10.1016/j.canlet.2022.215649. Epub 2022 Mar 18. PMID 35315341
- [Derived] Liu N, Zhang J, Yin M, Liu H, Zhang X, Li J, Yan B, Guo Y, Zhou J, Tao J, Hu S, Chen X, Peng C. Inhibition of xCT suppresses the efficacy of anti-PD-1/L1 melanoma treatment through exosomal PD-L1-induced macrophage M2 polarization. Mol Ther. 2021 Jul 7;29(7):2321-2334. doi: 10.1016/j.ymthe.2021.03.013. Epub 2021 Mar 17. PMID 33744468